CLINICAL TRIAL: NCT04012957
Title: A Phase 3, Multicenter, Multi-country, Open-label, Randomized, Active-controlled Clinical Trial to Evaluate the Efficacy and Safety of Desidustat Versus Darbepoetin for the Treatment of Anemia in Patients With Chronic Kidney Disease (CKD) Who Are Not on Dialysis
Brief Title: Desidustat in the Treatment of Anemia in CKD
Acronym: DREAM-ND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DESI.18.001
Record Dates: First submitted 2019-06-07; First posted 2019-07-09 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2020-07

CONDITIONS: Chronic Kidney Disease Stage 3; Anemia; Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5
Keywords: DREAM-ND
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — desidustat; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Darbepoetin Alfa Injection (Experimental): Randomly assigned to receive Darbepoetin in a 1:1 ratio for 24 weeks.
  Interventions: Drug: Darbepoetin Alfa
- Desidustat oral tablet (Active Comparator): Randomly assigned to receive Desidustat 100 mg in a 1:1 ratio for 24 weeks.
  Interventions: Drug: Desidustat Oral Tablet

INTERVENTIONS:
Drug: Desidustat Oral Tablet — Desidustat tablet
  Arms: Desidustat oral tablet
Drug: Darbepoetin Alfa — Darbepoetin injection
  Arms: Darbepoetin Alfa Injection

SUMMARY:
This is a phase III, multicenter, multi-country, open-label, randomized, active-controlled clinical trial to evaluate the efficacy and safety of Desidustat versus Darbepoetin for the treatment of anemia in patients with CKD who are not on dialysis. The study will be conducted over a period of up to 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Current clinical diagnosis of anemia due to CKD, baseline hemoglobin concentrations must be 7.0-10.0 g/dL (both inclusive) before the enrollment.
2. Ability to understand and give informed consent for participation.
3. Male or female patients diagnosed with CKD (stage III to V, not receiving dialysis) defined by estimated glomerular filtration rate (eGFR) using the CKD Epidemiology Collaboration (CKD-EPI) formula.
4. Male or female, 18 to 80 years of age.
5. Body weight > 40 kg.
6. Subjects not on dialysis and not expected to start dialysis during the study period.
7. Patients must not be treated with erythropoiesis-stimulating agent (ESA) therapy within 6 weeks prior to enrollment.
8. Estimated GFR ≥10 mL/min/1.73 m2.
9. Serum ferritin ≥100 ng/mL and/or Transferrin Saturation >20%.
10. No iron, folate or Vitamin B12 deficiency.
11. Females of childbearing potential, must agree to use one of the approved contraception methods, from screening until completion of the follow-up visit.

Exclusion Criteria:

1. Prior chronic hemodialysis or chronic peritoneal dialysis treatment.
2. Intravenous iron within 14 days prior to enrollment.
3. Prior exposure of rhEPO analogues less than 04 weeks.
4. Red blood cell transfusion within 8 weeks prior to enrollment.
5. History of previous or concurrent cancer.
6. Serologic status reflecting active hepatitis B or C infection or Human immunodeficiency virus (HIV) infection.
7. Active infection prior to enrollment.
8. History of renal transplant.
9. Major surgery within 90 days of the first day of study drug dosing, and minor surgery within 30 days of the first day of study drug dosing.
10. Unable to swallow tablets or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption such as; mal-absorption syndrome, resection of the small bowel or poorly controlled inflammatory bowel disease affecting the small intestine.
11. History of uncontrolled autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura (ITP) or thalassemia.
12. Presence or a history of bleeding disorders or clinical conditions (e.g. gastrointestinal [GI] bleeding or constitutional disorders) that may increase risk of life-threatening bleeding.
13. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
14. History of severe allergic or hypersensitivity to investigational products and its excipients.
15. Requires or is receiving anticoagulation with warfarin or equivalent vitamin K antagonists or other medications within 28 days of the first dose of study drug that in the investigator's opinion, could compromise patient safety.
16. Pregnant and breastfeeding women.
17. Current life-threatening illness, medical condition or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety.
18. Other laboratory abnormalities that, in the opinion of the investigator, would compromise the patient's safety or interfere with data interpretation.
19. Presence of other systemic disorders or diseases (e.g., respiratory, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or any other body system involvement) which, in the Investigator's opinion, could compromise the patient's safety.
20. History of significant alcoholism or drug abuse within the past 1 year. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco/nicotine products (more than 10 times per day).
21. History of difficulty with donating blood.
22. History or presence of any clinically significant ECG abnormalities during screening.
23. Participants who have participated in any drug research study other than the present trial within past 3 months.
24. Participants who have donated one unit (350 ml) of blood in the past 3 months or history of whole blood transfusion in last 120 days prior to enrollment.
25. History of chronic inflammatory disease (RA, Celiac disease, UC, Crohns disease, Systemic Lupus Erythematosus [SLE]).
26. In case of Diabetes mellitus patients, glycosylated haemoglobin (HbA1c) >9 %.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 24 weeks
  Change in Hb levels from baseline

SECONDARY OUTCOMES:
Hemoglobin Response | 24 weeks
  No. of subjects with Hb response
Hemoglobin target range | 24 weeks
  Time to achieve target range Hb level

CONTACTS AND LOCATIONS:
Overall Officials: DrDeven Parmar, MD, Study Director — Zydus Lifesciences Limited
Locations (31):
- India (31):
  - Sunrise Hospital, Vijayawada, Andhra Pradesh
  - HCG Hospital, Ahmedabad, Gujarat
  - Sangini Hospital, Ahmedabad, Gujarat
  - GSC Medical College and Research Centre, Ahmedabad, Gujarat
  - Thakershey Charitable trust Hospital, Ahmedabad, Gujarat
  - BAPS Pramukh Swami Hospital, Surat, Gujarat
  - Sterling Hospital, Vadodara, Gujarat
  - Dhiraj General Hospital, Vadodara, Gujarat
  - Sapthagiri Institute of Medical Sciences, Bangalore, Karnataka
  - Kasturba Medical College, Mangalore, Karnataka
  - Amrita Institute of Medical Science, Kochi, Kerala
  - Government Medical College, Kozhikode, Kerala
  - Mahatma Gandhi Mission Medical College & Hospital, Aurangabad, Maharashtra
  - Nav Sanjeevani Hospital (Sankalp Speciality Healthcare Pvt. Ltd), Nashik, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Bhaktivedanta Hospital and Research Institute, Thane, Maharashtra
  - Asian Institute Of Medical Sciences (AIMS) Hospital, Thane, Maharashtra
  - Max Super Specialty Hospital, New Delhi, National Capital Territory of Delhi
  - Fortis Hospital, Delhi, New Delhi
  - Apollo Hospital, Bhubaneswar, Odisha
  - Sardar Patel Medical College, Bikaner, Rajasthan
  - Sawai Man Singh (SMS) Medical College and Hospital, Jaipur, Rajasthan
  - Eternal Hospital, Jaipur, Rajasthan
  - Rukmani Birla Hospital, Jaipur, Rajasthan
  - Osmania General Hospital, Hyderabad, Telangana
  - Apollo Hospital, Hyderabad, Telangana
  - Nizams Institute of Medical Sciences, Hyderabad, Telangana
  - Heritage Hospitals Limited, Varanasi, Uttar Pradesh
  - Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
  - Medica Superspecialty Hospital, Kolkata, West Bangal
  - Peerless Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278